CLINICAL TRIAL: NCT04803968
Title: The Effect of Upper Extremity Endurance Training Applied in Addition to Lower Extremity Endurance Training on Functional Capacity and Pacemaker Functions in Heart Failure Patients With Implantable Cardioverter Defibrillator (ICD)
Brief Title: The Effect of Combined Upper and Lower Extremity Endurance Training in Patients With ICD
Acronym: ICD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hitit University (Other)
Collaborators: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ayşe Akdal, physiotherapist, Hitit University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 322
Record Dates: First submitted 2021-03-15; First posted 2021-03-18 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Heart Failure With Reduced Ejection Fraction
Keywords: Implantable cardiac defibrillator; Upper extremity endurance training; peak Oxygen consumption; upper extremity functional capacity

STUDY DESIGN:
Intervention Model Description: randomized controlled clinical trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Experimental): After the evaluations are completed, the participants will be randomly divided into two groups using a computer-assisted randomization program.
  The cardiac rehabilitation program will be a total of 30 sessions, 5 days a week x 6 weeks. All patients in the control and study groups will participate in the routine lower extremity bicycle ergometer training
  Interventions: Other: bicycle ergometer exercise
- intervention group (Experimental): The combined upper and lower extremity training group will participate in the arm ergometer exercise separately from the lower extremity training group.
  Interventions: Other: bicycle ergometer and arm ergometer exercise

INTERVENTIONS:
Other: bicycle ergometer and arm ergometer exercise — After the bicycle ergometer training is completed, there will be a 15-minute break for blood pressure measurement of the patients.
  Then the combined upper and lower extremity training group will participate in the arm ergometer exercise separately from the lower extremity training group.
  For this, the patient will sit upright in front of the height-adjustable arm ergometer stand (Lode Angio Arm Ergometer with Automat) with the fulcrum of the handle at shoulder height.
  The arm endurance training group will work for a total of 20 minutes, at 60% of the peak workload and at 50 rpm.
  Arms: intervention group
Other: bicycle ergometer exercise — All patients in the control and study groups will participate in the routine lower extremity bicycle ergometer training (Lode Corival Cpet Ergoline type: 960900 serial number: 20160094, Netherlands). The exercise protocol for the lower extremities will consist of a total of 40 minutes, including an 8-minute warm-up phase and an 8-minute cool-down phase. Exercise intensity, on the other hand, will be arranged as recommended in the European Society of Cardiology (ESC) 2020 guideline for chronic heart failure patients, at a workload corresponding to 70-80% of peak oxygen consumption (VO2peak), with a turnover rate of 60 cycles / min.
  Arms: control group

SUMMARY:
It was aimed to examine whether the arm endurance exercise training is effective in addition to the lower cycling training program in order to alleviate the negative functional results in heart failure patients with ICD.

DETAILED DESCRIPTION:
Pacemaker (permanent battery) is implanted in patients for many reasons. For reasons such as symptomatic bradycardia and AV block, a pacemaker with modes such as VVR and DDDR designed for pacing only when the pulse decreases can be implanted. At the same time, pacemakers can be implanted in VR-ICD, DR-ICD modes, which have the ability to recognize fatal rhythm problems such as Ventricular tachycardia (VT) / Ventricular Fibrillation (VF) and perform intracardiac defibrillation (ICD).

Pacemakers are positioned by opening a pocket under the patient's left pectoral muscle.Cables coming out of the battery (leads) are placed in the right ventricle, right atrium or coronary sinuses via active or passive fixation through the left subclavian vein. In the early period after pacemaker implantation, patients are warned to avoid movements that force the extremity on that side so that the leads and battery are affected by extremity movements and their positions and functions are not impaired.

Many pacemaker patients prolong this period too much (> 3 months), causing them to develop left extremity muscle-joint dysfunction. This situation can also affect the functional capacity of the patients.ICD pacemakers are larger in size than conventional pacemakers due to their functions, so they are placed in a larger pocket in the pectoral area.These patients are warned more strictly about coercive movements.

The aim of this study is to investigate the effect of arm ergometer endurance training on functional capacity and upper extremity function in heart failure patients with ICD included in cardiac rehabilitation program, and to examine the effect on battery and leads as safety parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of heart failure in the New York Heart Association (NYHA) class II-III, who have had at least 3 months past ICD implantation, and who did not have any complications at the last pacemaker control,
* Ejection fraction (EF) value ≤45%,
* The medicines used have not been changed for at least 3 months,
* Volunteering to participate in the research, being able to attend a 1-hour rehabilitation program every day of the week,
* To be clinically stable, to be under control if any accompanying comorbid conditions (such as hypertension, diabetes),
* Not having any orthopedic problems that may prevent him from exercising with his bicycle and arm ergometer,
* CPET, ambulatory blood pressure and rhythm monitoring, ECG and ECHO without any obstacle to exercise within the framework of TKD cardiology guidelines (such as moderate valve disease, hypertrophic cardiomyopathy, severe uncontrolled HT…).

Exclusion Criteria:

* Those with a history of shoulder injury (severe pain around the shoulder and inability to move, severe swelling around the shoulder, shoulder dislocation)
* Those with a history of shoulder surgery,
* Sequelae of a cerebrovascular accident with mastectomy or arm involvement on the affected side,
* Having decompensated heart failure,
* Having an obstacle to exercise within the framework of TSC (Turkish Society of Cardiology) cardiology guidelines in CPET, ambulatory blood pressure and rhythm monitoring, ECG and ECO (such as moderate valve disease, hypertrophic cardiomyopathy, severe uncontrolled HT ...)
* Having a history of ICD shock in the last 6 months,
* Having an active treated malignancy or a collagen tissue disease receiving systemic steroids
* Being unable to cooperate or adapt to exercise due to cerebrovascular disease or other reasons,
* Having a chronic kidney disease undergoing dialysis where the volume load is not stable.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Cardiorespiratory functional capacity | Through study completion, an average of 1 year
  Cardiopulmonary exercise test (CPET):
  It evaluates the aerobic capacity before the rehabilitation program and evaluates the responses to exercise and is used as the gold standard. A ramp bicycle ergometer test protocol will be applied for CPET. Parameters such as exercise duration, Watt, VO2, VCO2, blood pressure, heart rate, dyspnea, leg fatigue, general fatigue and effort perception according to the modified Borg scale, SaO2 will be saved at rest, AT (at anaerobic threshold), at peak level and at the end of the test in the recovery phase.
  At the end of the test, the reason for completing the test will be recorded. As one of the criteria for completing the test, attention will be paid to having the RER value of 1.05 and above. Results will be printed with 9 panel charts. (Gas analyzer; CORTEX METALYZER 3B Germany, bicycle; Lode Corival-cpet ERGOMETER, 12 channel ECG test system; Custo Cardio 200 BT system, Netherlands)
Arm ergometer endurance capacity | Through study completion, an average of 1 year
  The Lode Angio Arm Ergometer (with automatic stand, type: 917900 serial number:20160739, The Netherlands) device will be used for the arm ergometer test. It will start rotating the arm ergometer at 0 Watt (W) workload and at a speed of 60-75 rpm and will progress with a 10 W workload increase every 2 minutes. Modified Borg scores will be recorded for the patient's perception of arm fatigue and dyspnea before each workload increase. When the patient reaches one of the test termination criteria, the test will be terminated and the last achieved workload will be recorded as W and due to termination of the test.
6 minute pegboard and ring test | Through study completion, an average of 1 year
  Participants will sit in front of a board with two top pegs, two bottom pegs and 10 rings on top of it. The lower pegs will be placed at the participant's shoulder height, and the upper pegs will be placed in the hole 20 cm above the lower pegs. Within a 6-minute period, participants will be asked to move as many rings as possible from the lower pegs to the upper pegs.
  Before and after each test, blood pressure, heart rate, SpO2 (Veron, VRN-502 pulse oximeter), dyspnea and arm fatigue detection (modified borg scale) will be recorded.
  The test will be performed a second time after the first test is completed, after a 30-minute interval or after the relevant variables return to their initial values. If the patient wants to rest during the test, they will be allowed but the stopwatch will not be stopped. During the test, patients will be encouraged every minute. The result of the test is the total number of rings carried.
Handgrip | Through study completion, an average of 1 year
  The measurements will be made in three repetitions for the right and left sides, with the shoulder in the sitting position, the elbow in 90 ° flexion, and the forearm in neutral position (Smedley Digital Hand Dynamometer, Model: 12-0286, Baseline, Fabrication Enterprises Inc (FEI), USA). For statistical analysis, the best values of the right and left sides and the arithmetic means of both sides will be recorded.

SECONDARY OUTCOMES:
Quick DASH | Through study completion, an average of 1 year
  It is an abbreviation of the 30-item Quick-DASH questionnaire used to evaluate one or more musculoskeletal physical functions and symptoms of the upper extremity. It consists of 11 items. The results of the questionnaire will be evaluated on a 100 point scale and higher scores will indicate the presence of more disability.
The Minnesota Living with Heart Failure Questionnaire (MLHFQ) | Through study completion, an average of 1 year
  The MLHFQ consists of 21 items and measures three important dimensions (physical, socioeconomic and psychological) of quality of life in patients with heart failure. It is scored with a 6-point Likert scale graded as 0 (no effect / not valid, best score) -5 (severe impact, worst score) within an average of 5 minutes. It can be applied by itself or by an interviewer.
  The total score of the scale for 21 questions ranges from 0 to 105, and higher scores indicate a lower quality of life.
  The patients' quality of life will be evaluated with the "Minnesota Heart Failure Life Questionnaire", which measures the quality of life specific to heart failure. The Turkish validity and reliability of the questionnaire has been done.
General Practice Physical Activity Questionnaire (GPPAQ) | Through study completion, an average of 1 year
  The "General Practice Physical Activity Questionnaire" (GPPAQ), which was developed to evaluate the physical activity level of adults in primary care, consists of seven questions under three main headings. It is a scale that takes about 30-60 seconds to fill. In the first part of the scale, a question is asked about the mobility of the person in the workplace, while the second part is asked about the activities performed in the last seven days and how many hours per week. In the last part, there is a question that evaluates the normal walking speed of the person.

CONTACTS AND LOCATIONS:
Locations (1):
- Hitit University, Çorum, Turkey (Türkiye)